CLINICAL TRIAL: NCT05702814
Title: Validation of a Set of Potential Biomarkers Predictive of Bone Complications in Type 1 Gaucher Disease Patients
Brief Title: A Study Measuring Substances Potentially Indicating Bone Problems in Adults With Type 1 Gaucher Condition
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-669-5010
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Gaucher Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: GD1 with Low-normal Bone Disease: Participants with GD1 with low-normal bone disease whose samples are available for analysis in BSSA will be collected retrospectively up to approximately 5 years from diagnosis.
  Interventions: Other: No Intervention
- Group B: GD1 with Mild Bone Disease: Participants with GD1 with mild bone disease whose samples are available for analysis in BSSA will be collected retrospectively up to approximately 5 years from diagnosis.
  Interventions: Other: No Intervention
- Group C: GD1 with Severe Bone Disease: Participants with GD1 with severe bone disease whose samples are available for analysis in BSSA will be collected retrospectively up to approximately 5 years from diagnosis.
  Interventions: Other: No Intervention
- Group D: Healthy Participants: Healthy Participants whose samples are available for analysis in BSSA will be collected retrospectively up to approximately 5 years.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As this is an observational study, no intervention will be administered.

SUMMARY:
Substances in the body, so-called biomarkers, can help predict the severity of Gaucher disease (GD)-related bone problems in adults. The main aim of the study is to determine if certain biomarkers found in the body at the time of diagnosing GD can help predict the risk of bone problems after 4-5 years.

There is no treatment involved in this study. The study will review previously collected participants' data using a database. Data from both adults with type 1 Gaucher condition as well as healthy adults will be compared.

DETAILED DESCRIPTION:
This is a non-interventional and retrospective study of participants with GD1 and healthy participants whose data is available in the Aragon Health Systems Biobank (BSSA) from the date of diagnosis to 4-5 years after diagnosis. The main objective of this study is to validate the prognosis value of a set of potential biomarkers related to bone disease in participants with GD1.

The study will enroll approximately 120 participants, and it would be divided into 4 groups as given below:

* Group A: GD1 with Low-Normal Bone Disease
* Group B: GD1 with Mild Bone Disease
* Group C: GD1 with Severe Bone Disease
* Group D: Healthy Participants

This study will have a retrospective data collection from the date of diagnosis of GD1 until 4-5 years from diagnosis by using data available in BSSA.

This single-centre trial will be conducted in Spain. The overall time for data collection in this study will be approximately 9 months.

ELIGIBILITY:
For Participants with GD1:

Inclusion Criteria

* Participants with confirmed diagnosis of GD1.
* Determination of Glucocerebrosidase (GCase) blood activity at diagnosis of GD1.
* DNA analysis result demonstrating pathogenic variants in the Glucocerebrosidase gene (GBA1) gene.
* Available data of clinical state at diagnosis and at 4-5 years from diagnosis, including S-MRI, Dual energy x-ray absorptiometry (DXA), and GD1 severity scoring system (GD1-DS3) indexes (or data to calculate it).

Exclusion Criteria

• Evidence of hepatitis B, hepatitis C infection or other chronic infectious diseases.

For Healthy Volunteers

Exclusion Criteria

* Evidence of hepatitis B, hepatitis C infection or other chronic infectious diseases.
* Evidence of bone disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with GD1 and healthy participants in Spain.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Change in Biomarker Level in Participants with GD1 at 4-5 years From Diagnosis Assessed per Spanish-Magnetic Resonance Imaging (S-MRI) | Baseline up to approximately 4-5 years
  Areas like spine, pelvis, and femora will be evaluated and the MRI pattern will be ranged as normal=0, non-homogenous reticular pattern=1, non-homogenous mottled pattern= 2, non-homogenous diffuse pattern= 3, and homogenous pattern=4, and the presence of complications adds a value of 4. For each site, the maximum possible value assigned is 8, and the S-MRI is the sum of the score obtained at each site; thus, the S-MRI score ranges from 0 to 24.

SECONDARY OUTCOMES:
Change in Biomarker Level in Participants with GD1 at Diagnosis as Assessed per S-MRI | Baseline (At diagnosis prior to treatment start)
  Areas like spine, pelvis, and femora will be evaluated and the MRI pattern will be ranged as normal=0, non-homogenous reticular pattern=1, non-homogenous mottled pattern= 2, non-homogenous diffuse pattern= 3, and homogenous pattern=4, and the presence of complications adds a value of 4. For each site, the maximum possible value assigned is 8, and the S-MRI is the sum of the score obtained at each site; thus, the S-MRI score ranges from 0 to 24.
Change in Biomarker Level At Diagnosis And Severity Of Bone Disease At Diagnosis As Assessed Per S-MRI in Participants with GD1 and no Bone Disease in Healthy Volunteers | Baseline (At diagnosis prior to treatment start)
Change in Biomarker Level At Diagnosis And Severity Of Bone Disease At Diagnosis As Assessed Per DXA in Participants with GD1 and no Bone Disease in Healthy Volunteers | Baseline (At diagnosis prior to treatment start)
Change in Biomarker Level at Diagnosis as Assessed per Gaucher Disease Type 1 Severity Scoring System (GD1-DS3) Score in Participants with GD1 | Baseline (At diagnosis prior to treatment start)
  GD1-DS3 score ranges from 0 to a maximum of 19 for the disease domains bone (lytic lesions, AVN or pathological fractures, bone/joint pain, bone crisis, bone marrow infiltration, bone mineral density), hematology (thrombocytopenia, bleeding and anaemia) and visceral (splenomegaly, hepatomegaly, and Gaucher-related pulmonary disease). GD1-DS3 total score is a sum of the above three disease domain scores ranging from 0-3= borderline to mild disease, 3-6= moderate disease, 6-9= Marked disease, and +9=Severe disease.
Change in Biomarker Level at 4-5 years from Diagnosis as Assessed per GD1-DS3 Score in Participants with GD1 | Baseline to approximately 4-5 years
  GD1-DS3 score ranges from 0 to a maximum of 19 for the disease domains bone (lytic lesions, AVN or pathological fractures, bone/joint pain, bone crisis, bone marrow infiltration, bone mineral density), hematology (thrombocytopenia, bleeding and anaemia) and visceral (splenomegaly, hepatomegaly, and Gaucher-related pulmonary disease). GD1-DS3 total score is a sum of the above three disease domain scores ranging from 0-3= borderline to mild disease, 3-6= moderate disease, 6-9= Marked disease, and +9=Severe disease.
Comparison Between in lyso-Gb1, ChT, CCL18, and Study Biomarkers Levels in Participants with GD1 and Healthy Volunteers at Diagnosis | Baseline (At diagnosis prior to treatment start)
Comparison Between in lyso-Gb1, ChT, CCL18, and Study Biomarkers Levels in Participants with GD1 and Healthy Volunteers at 4-5 years at Diagnosis | Baseline to approximately 4-5 years
Change From Baseline in lyso-Gb1, ChT, CCL18, and Study Biomarkers Levels in Participants with GD1 and Healthy Volunteers at Diagnosis | Baseline (At diagnosis prior to treatment start)
Change From Baseline in lyso-Gb1, ChT, CCL18, and Study Biomarkers Levels in Participants with GD1 at years at Diagnosis | Baseline to approximately 4-5 years
Change From Baseline in Lumbar DXA Measurements: Bone Mineral Density (BMD), Z- score from Diagnosis | Baseline and up to approximately 4-5 years
  Bone mineral density of the lumbar spine would be measured by dual energy x-ray absorptiometry (DXA), and the results would be converted to Z-scores appropriate for age, sex, and race. The Z-score indicated the number of standard deviations away from a reference population in the same age range, race and with the same sex. A Z-score of 0 was equal to the mean. Negative numbers indicated values lower than the mean and positive numbers indicated values higher than the mean.
Change From Baseline in Lumbar DXA Measurements: Bone Mineral Density (BMD), T- score from Diagnosis | Baseline and up to approximately 4-5 years
  BMD T-score is the standard deviation of the difference between measured BMD and that of the healthy young adult "normal". The T-score scale was as follows: -1 and above=normal, -1 to -2.5=osteopenia (below normal and may lead to osteoporosis), and -2.5 and below=osteoporosis.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Fundación Española para el Estudio y Tratamiento de la Enfermedad de Gaucher (FEETEG), Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/